CLINICAL TRIAL: NCT01733342
Title: Single-center Randomized Trial for Comparison of Performance Between Domestic and Imported Chemoport
Acronym: SiCDIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Cheol Kim, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP2012-k
Record Dates: First submitted 2012-11-13; First posted 2012-11-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celsite (Active Comparator): patients received celsite chemoport implantation under local anesthesia
  Interventions: Device: Celsite chemoport implantation; Procedure: local anesthesia
- Humanport (Experimental): patients received Humanport chemoport implantation under local anesthesia
  Interventions: Procedure: local anesthesia; Device: Humanport chemoport implantation

INTERVENTIONS:
Device: Celsite chemoport implantation — Celsite chemoport implantation was done under local anesthesia, at anterior chest wall, under ultrasound guidance
  Arms: Celsite
Procedure: local anesthesia — chemoport implantation will be done under local anesthesia using lidocaine.
Device: Humanport chemoport implantation — Humanport chemoport implantation was done under local anesthesia, at anterior chest wall, under ultrasound guidance
  Arms: Humanport

SUMMARY:
To compare the performance of domestic chemoport and imported chemoport

DETAILED DESCRIPTION:
chemoport implantation was done by two investigator Chemoport type was randomly rendered. Domestic chemoport(Human port) and imported chemoport (Celsite) were used. chemoport function will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* patients who will receive chemotherapy via implantable port
* age >20 years
* expected life time > 6 months
* lab test (platelet>50K, PT INR <2.0)

Exclusion Criteria:

* performance status >2
* brain metastasis
* expected life time less than 6 months
* age less than 20 years
* active infection
* severe heart dysfunction
* recent myocardial infarct

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
function of chemoport | 6 months
  Whether or not chemoport function is intact will be assessed. Chemoport function will be rendered as intact when chemotherapeutic agent is well infused through the chemoport. Chemoport function will be rendered as not intact when chemotherapeutic agent could be infused through the chemoport.

SECONDARY OUTCOMES:
infection | 6 months
  If infection related with chemoport develop during 6 month follow-up, infection will be recorded.
Skin dehiscence | 6 months
  If skin dehiscence related with chemoport develop during 6 month follow-up, it will be recorded.
deep vein thrombosis | 6 months
  If deep vein thrombosis related with chemoport develop during 6 month follow-up, it will be recorded. Deep vein thrombosis can be develop in the jugular vein which is access route.
Fibrin sheath | 6 months
  If fibrin sheath around chemoport catheter develop during 6 month follow-up, it will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Cheol Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Niederhuber JE, Ensminger W, Gyves JW, Liepman M, Doan K, Cozzi E. Totally implanted venous and arterial access system to replace external catheters in cancer treatment. Surgery. 1982 Oct;92(4):706-12. PMID 7123491
- [Background] Ahn SJ, Kim HC, Chung JW, An SB, Yin YH, Jae HJ, Park JH. Ultrasound and fluoroscopy-guided placement of central venous ports via internal jugular vein: retrospective analysis of 1254 port implantations at a single center. Korean J Radiol. 2012 May-Jun;13(3):314-23. doi: 10.3348/kjr.2012.13.3.314. Epub 2012 Apr 17. PMID 22563269
- [Background] Teichgraber UK, Kausche S, Nagel SN, Gebauer B. Outcome analysis in 3,160 implantations of radiologically guided placements of totally implantable central venous port systems. Eur Radiol. 2011 Jun;21(6):1224-32. doi: 10.1007/s00330-010-2045-7. Epub 2011 Jan 5. PMID 21207035
- [Background] Teichgraber UK, Kausche S, Nagel SN. Evaluation of radiologically implanted central venous port systems explanted due to complications. J Vasc Access. 2011 Oct-Dec;12(4):306-12. doi: 10.5301/JVA.2011.7739. PMID 21534232
- [Background] Biffi R, de Braud F, Orsi F, Pozzi S, Mauri S, Goldhirsch A, Nole F, Andreoni B. Totally implantable central venous access ports for long-term chemotherapy. A prospective study analyzing complications and costs of 333 devices with a minimum follow-up of 180 days. Ann Oncol. 1998 Jul;9(7):767-73. doi: 10.1023/a:1008392423469. PMID 9739444